CLINICAL TRIAL: NCT07017842
Title: PREDICT-H Study: Prospective Research on Essential Determinants Influencing Complication Trends in Hypospadias - a Landmark Prospective Multicenter Cohort Study Aimed at Improving Outcome Prediction in Hypospadias Surgery
Acronym: PREDICT-H
Status: Recruiting | Type: Observational
Sponsor: Sidra Medicine (Other)
Responsible Party: Principal Investigator, Tariq Abbas, Consultant Pediatric Urologist, Sidra Medicine
Other Study IDs: SDR600058
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypospadias (Age 1-12 years old): This study includes a single prospective observational cohort of male pediatric patients aged 1 to 12 years undergoing primary surgical repair for hypospadias at participating tertiary pediatric urology centers. No experimental interventions are assigned by the study; instead, patients receive standard-of-care surgical techniques as determined by their treating surgeons. Detailed preoperative anatomical assessments and surgical procedure documentation are collected to evaluate the impact of anatomical variables and surgical approaches on postoperative complication rates. Subgroup analyses will be performed based on hypospadias severity (distal, midpenile, proximal) and the surgical technique utilized.

SUMMARY:
Hypospadias is a common congenital anomaly with complex anatomy that influences surgical outcomes. Despite numerous surgical techniques, a lack of standardized preoperative assessment protocols and consensus on anatomical risk factors limits prediction of complications. This study aims to systematically evaluate key anatomical features identified in previous meta-analyses-such as urethral plate width and length, glans size, chordee severity, meatal position, and others-in a large, prospective multicenter cohort. The ultimate goal is to develop and validate an objective nomogram predicting the risk of postoperative complications, enabling individualized surgical planning and improved patient counseling.

ELIGIBILITY:
* Inclusion Criteria:

Male patients aged 1 to 12 years

Diagnosed with hypospadias (distal, midpenile, proximal)

Undergoing primary surgical repair

Parent/legal guardian consent obtained

* Exclusion Criteria:

Prior hypospadias or penile surgery (revision cases)

Major associated genital anomalies (e.g., ambiguous genitalia, severe DSD)

Refusal of consent or inability to complete follow-up

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Study Population: Male patients aged 1 to 12 years with diagnosed distal, midpenile, or proximal hypospadias scheduled for primary surgical repair will be enrolled. Exclusion criteria include prior hypospadias or penile surgery, major genital anomalies (e.g., ambiguous genitalia, severe DSD), inability or refusal to consent, or incomplete follow-up. Patients will be recruited from multiple tertiary pediatric urology centers. Informed consent will be obtained from parents or legal guardians. All participants will be followed for a minimum of 6 months postoperatively to assess surgical outcomes and complications.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: | minimum 6 months post-surgery
  Composite rate of postoperative complications within 6 months, including: urethrocutaneous fistula, meatal stenosis, urethral stricture, recurrent chordee, wound infection requiring treatment, and need for surgical revision.

SECONDARY OUTCOMES:
Individual Complication Rates Following Hypospadias Repair | At 1 month, 3 months, and a minimum of 6 months post-surgery; optional assessment at 12 months and last clinic visit
  The frequency of specific postoperative complications-including urethrocutaneous fistula, meatal stenosis, urethral stricture, recurrent chordee, wound infection, and need for surgical revision-will be assessed in patients undergoing primary hypospadias repair.
Cosmetic and Functional Outcomes After Hypospadias Surgery | At 1 month, 3 months, and a minimum of 6 months post-surgery; optional assessment at 12 months or last clinic visit
  Cosmetic appearance and functional urinary outcomes will be evaluated using validated scoring systems and satisfaction surveys completed by surgeons and parents at follow-up visits scheduled at 1, 3, and 6 months post-surgery. A minimum follow-up of 6 months is required for all patients, with an optional assessment at 12 months for long-term outcome validation.
Correlation Between Preoperative Anatomical Variables and Specific Postoperative Complications | Based on data collected during a minimum 6 months after surgery
  Statistical analyses will evaluate associations between preoperative anatomical measurements and individual postoperative complications. Data collection and follow-up for these analyses require a minimum postoperative period of 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidra Medicine, Doha, Baladīyat ad Dawḩah, Qatar

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including anatomical measurements, surgical details, and postoperative outcomes, will be made available to qualified researchers upon reasonable request following publication of the primary study results. Data sharing will comply with all applicable privacy regulations and institutional policies to ensure participant confidentiality. Requests will be reviewed by the study steering committee, and data will be shared via a secure platform after completion of a data use agreement.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Merriman LS, Arlen AM, Broecker BH, Smith EA, Kirsch AJ, Elmore JM. The GMS hypospadias score: assessment of inter-observer reliability and correlation with post-operative complications. J Pediatr Urol. 2013 Dec;9(6 Pt A):707-12. doi: 10.1016/j.jpurol.2013.04.006. Epub 2013 May 15. PMID 23683961
- [Background] Abbas TO, Khalil IA, Hatem M, Boyko A, Zorkin S. Plate Objective Scoring Tool (POST) in distal hypospadias: Correlation with post-repair complications. J Pediatr Urol. 2024 Apr;20(2):238.e1-238.e6. doi: 10.1016/j.jpurol.2023.11.022. Epub 2023 Nov 25. PMID 38071112
- [Background] Baray SB, Abdelmoniem M, Mahmud S, Kabir S, Faisal MAA, Chowdhury MEH, Abbas TO. Automated measurement of penile curvature using deep learning-based novel quantification method. Front Pediatr. 2023 Apr 17;11:1149318. doi: 10.3389/fped.2023.1149318. eCollection 2023. PMID 37138577
- [Background] Abbas TO, Vallasciani S, Elawad A, Elifranji M, Leslie B, Elkadhi A, Pippi Salle JL. Plate Objective Scoring Tool (POST); An objective methodology for the assessment of urethral plate in distal hypospadias. J Pediatr Urol. 2020 Oct;16(5):675-682. doi: 10.1016/j.jpurol.2020.07.043. Epub 2020 Aug 5. PMID 32830060
- [Background] Abbas TO. An objective hypospadias classification system. J Pediatr Urol. 2022 Aug;18(4):481.e1-481.e8. doi: 10.1016/j.jpurol.2022.05.001. Epub 2022 May 11. PMID 35644790
- See also: Hypospadias Registry — https://www.sidra.org/research/clinical-research/clinical-research-at-sidra-medicine/real-time-international-collaborative-hypospadias-database-rich/